CLINICAL TRIAL: NCT01610414
Title: Observer-blind Study to Evaluate Efficacy, Safety, and Immunogenicity of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A
Brief Title: Study to Evaluate Efficacy, Safety, and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Herpes Zoster Vaccine GSK1437173A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 115523; 2012-000138-20 (EudraCT Number)
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Herpes Zoster
Keywords: Observer-blind; Efficacy; Immunogenicity; Vaccination; Safety; Adult autologous haematopoietic cell transplant recipients; Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- GSK1437173A Group (Experimental): Subjects received 2 doses of the candidate HZ vaccine GSK 1437173A, administered intramuscularly (IM) in deltoid region of non-dominant arm, according to a 0, 1 Month schedule.
  Interventions: Biological: Herpes Zoster vaccine GSK1437173A
- Placebo Group (Placebo Comparator): Subjects received 2 doses of placebo (saline solution), administered intramuscularly (IM) in deltoid region of non-dominant arm, according to a 0, 1 Month schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Herpes Zoster vaccine GSK1437173A — 2 doses administered intramuscularly (IM) in deltoid region of non-dominant arm
  Arms: GSK1437173A Group
Biological: Placebo — 2 doses administered IM in deltoid region of non-dominant arm
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the efficacy of GSK Biologicals' vaccine GSK1437173A in the prevention of Herpes zoster (HZ) in autologous haematopoietic cell transplant recipients 18 years of age and older. To this end, the study will evaluate vaccine efficacy (VE) of the GSK1437173A vaccine, administered on a 2-dose schedule, compared to placebo in reducing the risk of developing HZ in this population.

ELIGIBILITY:
Inclusion Criteria:

Study entry (enrollment) occurs at the Pre-vaccination visit.

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* A male or female aged 18 years or older at the time of study entry.
* Has undergone or will undergo autologous HCT within 50-70 days prior to the first vaccination with the study vaccine/placebo, and there are no plans for additional HCTs.
* Female subjects of non-childbearing potential may be enrolled in the study. For this study population, non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.

OR Female subjects of childbearing potential may be enrolled in the study, if the subject has practiced adequate contraception for 30 days prior to vaccination with the study vaccine/placebo, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period and for 12 months after completion of the vaccination series (i.e., until Month 13).

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine/placebo, or planned use during the study period. However, the investigational use of a registered or non-registered product to treat the subject's underlying disease for which the HCT was undertaken, or a complication of the underlying disease, is allowed.
* Previous vaccination against HZ or varicella within the 12 months preceding the first dose of study vaccine/placebo.
* Planned administration during the study of a HZ vaccine other than the study vaccine.
* Occurrence of a varicella or HZ episode by clinical history within the 12 months preceding the first dose of study vaccine/placebo.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine or study material and equipment.
* Prophylactic antiviral therapy with activity against Varicella Zoster Virus (VZV) expected to last more than 6 months after transplantation.
* Administration and/or planned administration of a vaccine not foreseen by the study protocol between HCT and 30 days after the last dose of study vaccine/placebo. However, licensed non-replicating vaccines may be administered up to 8 days prior to dose 1and/or 2, and/or at least 14 days after any dose of study vaccine/placebo.
* HIV infection by clinical history.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions (if of childbearing potential) before Month 13 (i.e., one year after the last dose of study vaccine/placebo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1877 (Actual)
Dates: Start 2012-07-13 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (146):
- United States (19):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Westwood, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Minneota, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Marshfield, Wisconsin
- Australia (9):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Waratah, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, East Melbourne, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Parkville, Victoria
- Belgium (8):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Jette
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- GSK Investigational Site, Sofia, Bulgaria
- Canada (6):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- Czechia (3):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- GSK Investigational Site, Tallinn, Estonia
- Finland (3):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (7):
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Rouen
- Germany (11):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Bayreuth, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Eschweiler, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Tuenmen
- Israel (2):
  - GSK Investigational Site, Hafia
  - GSK Investigational Site, Jerusalem
- Italy (8):
  - GSK Investigational Site, Cona (FE), Emilia-Romagna
  - GSK Investigational Site, Meldola (FC), Emilia-Romagna
  - GSK Investigational Site, Ravenna, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Aviano (PN), Friuli Venezia Giulia
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Novara, Piedmont
- Japan (10):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Malaysia (2):
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kuala Selangor
- GSK Investigational Site, Leiden, Netherlands
- New Zealand (3):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Grafton
  - GSK Investigational Site, Wellington
- GSK Investigational Site, Panama City, Panama
- Poland (3):
  - GSK Investigational Site, Gliwice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Warsaw
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Târgu Mureş
- Russia (5):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Petrozavodsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, St'Petersburg
- South Africa (4):
  - GSK Investigational Site, Parktown, Gauteng
  - GSK Investigational Site, Plumstead, Western Province
  - GSK Investigational Site, Groenkloof
  - GSK Investigational Site, Moreleta Park, Pretoria
- South Korea (6):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jellanamdo
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Kyunggi-do
  - GSK Investigational Site, Seoul
- Spain (14):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Badalona/Barcelona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, León
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Murcia (El Palmar)
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Valencia
- Taiwan (3):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taoyuan Hsien
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Izmir
- United Kingdom (7):
  - GSK Investigational Site, Airdrie, Lanarkshire
  - GSK Investigational Site, Swindon, Wiltshire
  - GSK Investigational Site, Bournemouth
  - GSK Investigational Site, Cottingham
  - GSK Investigational Site, Headington, Oxford
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, Manchester

REFERENCES:
- [Derived] Matthews S, Curran D, Sabater Cabrera E, Boutry C, Lecrenier N, Cunningham AL, Schmader K. An Analysis of How Herpes Zoster Pain Affects Health-related Quality of Life of Placebo Patients From 3 Randomized Phase III Studies. Clin J Pain. 2023 Aug 1;39(8):386-393. doi: 10.1097/AJP.0000000000001129. PMID 37166199
- [Derived] Kim JH, Johnson R, Kovac M, Cunningham AL, Amakrane M, Sullivan KM, Dagnew AF, Curran D, Schuind A. Adjuvanted recombinant zoster vaccine decreases herpes zoster-associated pain and the use of pain medication across 3 randomized, placebo-controlled trials. Pain. 2023 Apr 1;164(4):741-748. doi: 10.1097/j.pain.0000000000002760. Epub 2022 Aug 19. PMID 36066965
- [Derived] Curran D, Matthews S, Rowley SD, Young JH, Bastidas A, Anagnostopoulos A, Barista I, Chandrasekar PH, Dickinson M, El Idrissi M, Heras I, Milliken ST, Monserrat Coll J, Navarro Matilla MB, Oostvogels L, Piatkowska-Jakubas B, Quiel D, Sabry W, Schwartz S, Selleslag DLD, Sullivan KM, Theunissen K, Yegin ZA, Yeh SP, Zaja F, Szer J; ZOE-HSCT Study group collaborators. Recombinant Zoster Vaccine Significantly Reduces the Impact on Quality of Life Caused by Herpes Zoster in Adult Autologous Hematopoietic Stem Cell Transplant Recipients: A Randomized Placebo-Controlled Trial (ZOE-HSCT). Biol Blood Marrow Transplant. 2019 Dec;25(12):2474-2481. doi: 10.1016/j.bbmt.2019.07.036. Epub 2019 Aug 5. PMID 31394276
- [Derived] Bastidas A, de la Serna J, El Idrissi M, Oostvogels L, Quittet P, Lopez-Jimenez J, Vural F, Pohlreich D, Zuckerman T, Issa NC, Gaidano G, Lee JJ, Abhyankar S, Solano C, Perez de Oteyza J, Satlin MJ, Schwartz S, Campins M, Rocci A, Vallejo Llamas C, Lee DG, Tan SM, Johnston AM, Grigg A, Boeckh MJ, Campora L, Lopez-Fauqued M, Heineman TC, Stadtmauer EA, Sullivan KM; ZOE-HSCT Study Group Collaborators. Effect of Recombinant Zoster Vaccine on Incidence of Herpes Zoster After Autologous Stem Cell Transplantation: A Randomized Clinical Trial. JAMA. 2019 Jul 9;322(2):123-133. doi: 10.1001/jama.2019.9053. PMID 31287523

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some of the enrolled subjects were allocated subject numbers, but were not administered all doses of study vaccine, hence they did not start the study.
Groups:
- GSK1437173A Group: Subjects received 2 doses of the candidate HZ vaccine GSK1437173A, administered intramuscularly (IM) in deltoid region of the non-dominant arm, according to a 0, 1-2-Months schedule.
- Placebo Group: Subjects received 2 doses of placebo (saline solution), administered intramuscularly (IM) in deltoid region of the non-dominant arm, according to a 0, 1-2-Months schedule.
Period: Study Start - Month 13
Arm/Group | GSK1437173A Group | Placebo Group
Started | 922 | 924
Completed | 807 | 795
Not Completed | 115 | 129
Not completed — Serious Adverse Event | 65 | 67
Not completed — Adverse Event | 14 | 14
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 23 | 30
Not completed — Migrated/moved from study area | 2 | 4
Not completed — Lost to Follow-up | 4 | 6
Not completed — Suspected HZ episode | 1 | 3
Not completed — Other reasons for withdrawal | 3 | 4
Period: Month 13 - Month 25
Arm/Group | GSK1437173A Group | Placebo Group
Started | 922 | 924
Completed | 857 | 854
Not Completed | 65 | 70
Not completed — Serious Adverse Event | 35 | 38
Not completed — Adverse Event | 8 | 4
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Migrated/moved from study area | 4 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 5 | 9
Not completed — Other reasons for withdrawal | 6 | 7
Period: After Month 25
Arm/Group | GSK1437173A Group | Placebo Group
Started | 922 | 924
Completed | 874 | 871
Not Completed | 48 | 53
Not completed — Study end not reached | 48 | 53

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A Group | Placebo Group | Total
Number analyzed (Participants) | 922 | 924 | 1846
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (11.7) | 55.1 (11.4) | 55.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 342 | 346 | 688
  Male | 580 | 578 | 1158
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage/African American | 15 | 25 | 40
  Geographic ancestry: American Indian or Alaskan Native | 2 | 0 | 2
  Geographic ancestry: Asian - Central/South Asian Heritage | 6 | 5 | 11
  Geographic ancestry: Asian - East Asian Heritage | 83 | 91 | 174
  Geographic ancestry: Asian - Japanese Heritage | 43 | 38 | 81
  Geographic ancestry: Asian - South East Asian Heritage | 18 | 16 | 34
  Geographic ancestry: White - Arabic/North African Heritage | 9 | 12 | 21
  Geographic ancestry: White - Caucasian/European Heritage | 715 | 712 | 1427
  Geographic ancestry: Mixed Origin | 31 | 25 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Confirmed Herpes Zoster (HZ) Episode
Description: A suspected case of HZ was defined as (1) a new rash characteristic of HZ (e.g., unilateral, dermatomal and accompanied by pain broadly defined to include allodynia, pruritus or other sensations), or a vesicular rash suggestive of VZV infection regardless of the distribution, and no alternative diagnosis; or (2) a clinical presentation (symptoms and/or signs) and specific laboratory findings* suggestive of VZV infection in the absence of characteristic HZ or VZV rash.
  A suspected case of HZ was confirmed either: by Polymerase Chain Reaction (PCR) or by the HZ Ascertainment Committee (HZAC), consisting of physicians with HZ expertise.
Time Frame: From Month 0 until the cut-off date for final analysis (median follow-up was of 21 months)
Population: The analysis was performed on the modified Total Vaccinated Cohort, which excluded subjects from the Total Vaccinated Cohort analysis who were not administered with the second vaccination or who received vaccine doses/or replacement not on the same group or who developed a confirmed case of HZ prior to 1 month after the second vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 870 | 851
Participants | 49 | 135
Statistical Analysis 1: Comparison: GSK1437173A Group vs Placebo Group; Vaccine efficacy (VE) was evaluated in the prevention of Herpes Zoster (HZ) in autologous haematopoietic stem cell transplant (HCT) recipients 18 years of agee and older; Test type: Superiority — Criterion: The lower limit (LL) of the 95% confidence interval (CI) for overall HZ vaccine efficacy was above 0%; p < 0.0001, Poisson method; Vaccine efficacy = 68.17, 95% CI 2-sided [55.56 to 77.53]

2. Secondary Outcome: Duration of 'Worst' HZ-associated Pain
Description: Duration of HZ-associated pain rated as 3 or greater on the 'worst pain' Zoster Brief Pain Inventory (ZBPI) question, following the onset of a confirmed HZ rash over the entire pain reporting period in subjects with confirmed HZ; presented as T (day) [=the sum of follow-up period (for subjects without severe worst pain T is 1, for subjects with severe worst pain T is the duration of severe worst pain) expressed in days].
Time Frame: From Month 0 until study end (4 years approximately), from the onset of a confirmed HZ rash over the entire pain reporting period
Population: The analysis was performed on the modified Total Vaccinated Cohort, which excluded subjects from the Total Vaccinated Cohort analysis, who developed a confirmed case of HZ prior to 1 month after the second vaccination.
Measure: Number; unit: T (day)
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 49 | 135
T (day) | 892.0 | 6275.0

3. Secondary Outcome: Number of Subjects With Confirmed HZ-associated Complications
Description: This analysis excluded complications that were linked to a confirmed HZ case that occurred after the start of the relapse treatment.
Time Frame: From Month 0 until the cut-off date for final analysis (median follow-up was of 21 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 870 | 851
Participants | 3 | 13

4. Secondary Outcome: Number of Subjects With Postherpetic Neuralgia (PHN)
Description: This analysis excluded PHN episodes that were linked to a confirmed HZ case that occurred after the start of the relapse treatment.
Time Frame: From Month 0 until study end (21 months median follow-up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 870 | 851
Participants | 1 | 9

5. Secondary Outcome: Antigen-glycoprotein E (gE) Antibody Concentrations in a Sub-cohort of Subjects
Description: Anti-gE antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL). The seropositivity cut-off value was greater than or equal to (≥) 97 mIU/mL.
Time Frame: At Months 0, 1, 2, 13 and 25
Population: The analysis was performed on the adapted According-to-Protocol (ATP) cohort for humoral immunogenicity, which included data from the ATP cohorts for humoral immunogenicity at Months 0,1,2,13 and 25. The ATP cohort for humoral immunogenicity included all subjects from humoral immunogenicity sub-cohort in ATP cohort for analysis of immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 82 | 76
mIU/mL
  Anti-gE, Month 0 | 762.8 [568.6 to 1023.5] | 555.0 [404.3 to 761.8]
  Anti-gE, Month 1: number analyzed (Participants) | 78 | 71
  Anti-gE, Month 1 | 1844.2 [1282.2 to 2652.4] | 556.6 [407.3 to 760.6]
  Anti-gE, Month 2 | 12753.2 [7973.0 to 20399.4] | 443.8 [330.8 to 595.4]
  Anti-gE, Month 13: number analyzed (Participants) | 54 | 45
  Anti-gE, Month 13 | 3183.8 [1869.8 to 5421.2] | 503.6 [307.8 to 824.1]
  Anti-gE, Month 25: number analyzed (Participants) | 39 | 28
  Anti-gE, Month 25 | 2819.0 [1387.1 to 5729.1] | 527.0 [274.3 to 1012.6]

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with respect to the vaccine actually administered, who had filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 901 | 892
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 896 | 890
  Any Pain, Dose 1 | 688 | 56
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 896 | 890
  Grade 3 Pain, Dose 1 | 59 | 3
  Any Redness, Dose 1: number analyzed (Participants) | 896 | 890
  Any Redness, Dose 1 | 187 | 5
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 896 | 890
  Grade 3 Redness, Dose 1 | 7 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 896 | 890
  Any Swelling, Dose 1 | 101 | 7
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 896 | 890
  Grade 3 Swelling, Dose 1 | 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 840 | 834
  Any Pain, Dose 2 | 638 | 45
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 840 | 834
  Grade 3 Pain, Dose 2 | 63 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 840 | 834
  Any Redness, Dose 2 | 231 | 4
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 840 | 834
  Grade 3 Redness, Dose 2 | 24 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 840 | 834
  Any Swelling, Dose 2 | 132 | 3
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 840 | 834
  Grade 3 Swelling, Dose 2 | 12 | 0
  Any Pain, Across doses | 756 | 83
  Grade 3 Pain, Across doses | 99 | 3
  Any Redness, Across doses | 301 | 9
  Grade 3 Redness, Across doses | 28 | 0
  Any Swelling, Across doses | 168 | 9
  Grade 3 Swelling, Across doses | 13 | 0

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, myalgia, shivering and fever [defined as axillary/tympanic temperature equal to or above 37.5 degrees Celsius (°C) or rectal temperature equal to or above 38.0 °C]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 901 | 894
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 896 | 892
  Any Fatigue, Dose 1 | 356 | 282
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 896 | 892
  Grade 3 Fatigue, Dose 1 | 30 | 16
  Related Fatigue, Dose 1: number analyzed (Participants) | 896 | 892
  Related Fatigue, Dose 1 | 124 | 55
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 896 | 892
  Any Gastrointestinal, Dose 1 | 150 | 134
  Grade 3 Gastrointestinal, Dose 1: number analyzed (Participants) | 896 | 892
  Grade 3 Gastrointestinal, Dose 1 | 6 | 7
  Related Gastrointestinal, Dose 1: number analyzed (Participants) | 896 | 892
  Related Gastrointestinal, Dose 1 | 41 | 22
  Any Headache, Dose 1: number analyzed (Participants) | 896 | 892
  Any Headache, Dose 1 | 156 | 121
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 896 | 892
  Grade 3 Headache, Dose 1 | 2 | 3
  Related Headache, Dose 1: number analyzed (Participants) | 896 | 892
  Related Headache, Dose 1 | 51 | 32
  Any Myalgia, Dose 1: number analyzed (Participants) | 896 | 892
  Any Myalgia, Dose 1 | 340 | 170
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 896 | 892
  Grade 3 Myalgia, Dose 1 | 22 | 11
  Related Myalgia, Dose 1: number analyzed (Participants) | 896 | 892
  Related Myalgia, Dose 1 | 170 | 50
  Any Shivering, Dose 1: number analyzed (Participants) | 896 | 892
  Any Shivering, Dose 1 | 116 | 73
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 896 | 892
  Grade 3 Shivering, Dose 1 | 6 | 6
  Related Shivering, Dose 1: number analyzed (Participants) | 896 | 892
  Related Shivering, Dose 1 | 56 | 27
  Any Temperature, Dose 1: number analyzed (Participants) | 896 | 892
  Any Temperature, Dose 1 | 60 | 28
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 896 | 892
  Grade 3 Temperature, Dose 1 | 1 | 0
  Related Temperature, Dose 1: number analyzed (Participants) | 896 | 892
  Related Temperature, Dose 1 | 27 | 7
  Any Fatigue, Dose 2: number analyzed (Participants) | 836 | 835
  Any Fatigue, Dose 2 | 395 | 212
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 836 | 835
  Grade 3 Fatigue, Dose 2 | 48 | 20
  Related Fatigue, Dose 2: number analyzed (Participants) | 836 | 835
  Related Fatigue, Dose 2 | 153 | 41
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 836 | 835
  Any Gastrointestinal, Dose 2 | 142 | 98
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 836 | 835
  Grade 3 Gastrointestinal, Dose 2 | 13 | 12
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 836 | 835
  Related Gastrointestinal, Dose 2 | 51 | 13
  Any Headache, Dose 2: number analyzed (Participants) | 836 | 835
  Any Headache, Dose 2 | 232 | 88
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 836 | 835
  Grade 3 Headache, Dose 2 | 24 | 8
  Related Any Headache, Dose 2: number analyzed (Participants) | 836 | 835
  Related Any Headache, Dose 2 | 95 | 20
  Any Myalgia, Dose 2: number analyzed (Participants) | 836 | 835
  Any Myalgia, Dose 2 | 374 | 153
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 836 | 835
  Grade 3 Myalgia, Dose 2 | 42 | 9
  Related Myalgia, Dose 2: number analyzed (Participants) | 836 | 835
  Related Myalgia, Dose 2 | 208 | 47
  Any Shivering, Dose 2: number analyzed (Participants) | 836 | 835
  Any Shivering, Dose 2 | 185 | 59
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 836 | 835
  Grade 3 Shivering, Dose 2 | 29 | 1
  Related Shivering, Dose 2: number analyzed (Participants) | 836 | 835
  Related Shivering, Dose 2 | 102 | 16
  Any Temperature, Dose 2: number analyzed (Participants) | 836 | 835
  Any Temperature, Dose 2 | 150 | 28
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 836 | 835
  Grade 3 Temperature, Dose 2 | 2 | 1
  Related Temperature, Dose 2: number analyzed (Participants) | 836 | 835
  Related Temperature, Dose 2 | 8 | 8
  Any Fatigue, Across doses | 508 | 340
  Grade 3 Fatigue, Across doses | 66 | 31
  Related Fatigue, Across doses | 210 | 79
  Any Gastrointestinal, Across doses | 238 | 183
  Grade 3 Gastrointestinal, Across doses | 18 | 17
  Related Gastrointestinal, Across doses | 79 | 30
  Any Headache, Across doses | 302 | 166
  Grade 3 Headache, Across doses | 26 | 10
  Related Headache, Across doses | 123 | 46
  Any Myalgia, Across doses | 484 | 234
  Grade 3 Myalgia, Across doses | 56 | 19
  Related Myalgia, Across doses | 279 | 83
  Any Shivering, Across doses | 237 | 115
  Grade 3 Shivering, Across doses | 35 | 7
  Related Shivering, Across doses | 131 | 38
  Any Temperature, Across doses | 183 | 50
  Grade 3 Temperature, Across doses | 3 | 1
  Related Temperature, Across doses | 101 | 15

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with respect to the vaccine actually administered.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 922 | 924
Participants
  Any AE(s) | 360 | 353
  Grade 3 AE(s) | 60 | 47
  Related AE(s) | 31 | 23

9. Secondary Outcome: Number of Subjects With Any and Related Potential Immune Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Month 0 up to 365 days post last vaccination
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 922 | 924
Participants
  Any pIMDs | 13 | 8
  Related pIMDs | 3 | 0

10. Secondary Outcome: Number of Subjects With Any Relapse
Description: Relapse was defined as the occurrence of the underlying malignancy or disease for which the HCT was undertaken.
Time Frame: From Month 0 until study end (approximate median of 29 months follow-up - minimum 1 year and maximum 4 years)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 922 | 924
Participants | 239 | 253

11. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) and Related SAEs to GSK Study Vaccine/Placebo
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject. This enpoint also presents SAES related to the GSK study vaccine/placebo.
Time Frame: From Month 0 until 365 days post last vaccination (approximate median of 29 months follow-up - minimum 1 year and maximum 4 years)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 922 | 924
Participants
  Any SAEs, up to Month 13 | 263 | 241
  Related SAEs, up to Month 13 | 3 | 4
  Any SAEs, up to Study End | 329 | 310

12. Secondary Outcome: Number of Subjects With Fatal SAEs and SAEs Related to Study Participation or to a GSK Concomitant Medication or Vaccination
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject. This endpoint presents fatal SAEs and SAEs related to study participation or to a concurrent GSK medication/vaccine.
Time Frame: From the Pre-vaccination visit (Up to 110 days prior Month 0) until study end (approximate median of 29 months follow-up minimum 1 year and maximum 4 years)
Population: The analysis was performed on the Total Enrolled Cohort.
Measure: Count of Participants; unit: Participants
Groups:
- No Group: Subjects who were not assigned to any group (subjects from pre-vaccination visit).
Arm/Group | GSK1437173A Group | Placebo Group | No Group
Number analyzed (Participants) | 932 | 933 | 3
Participants
  Fatal SAEs | 118 | 124 | 0
  Related SAEs | 37 | 43 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited adverse events (AEs): during the 30-day (Days 0-29) post-vaccination period; SAEs: during the entire study period, up to 365 days post last vaccination (4 years approximately).
Arm/Group | GSK1437173A Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 118/922 | 124/924
Serious Adverse Events (participants affected / at risk) | 329/922 | 310/924
Other Adverse Events (participants affected / at risk) | 813/922 | 485/924
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=922) | Placebo Group (N=924)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (16) | 12 (13)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Haematotympanum (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 2 (2)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 2 (2) | 2 (2)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 3 (3)
Hernia (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 10 (11) | 8 (9)
Sudden death (General disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Chronic graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease (Immune system disorders) | 6 (6) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease in skin (Immune system disorders) | 1 (1) | 2 (2)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 3 (3) | 3 (4)
Bacterial infection (Infections and infestations) | 1 (1) | 2 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 6 (6)
Bronchopulmonary aspergillosis (Infections and infestations) | 4 (4) | 2 (2)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 4 (4)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 3 (3)
Device related infection (Infections and infestations) | 2 (2) | 3 (3)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1)
Epstein-barr viraemia (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 2 (2)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Febrile infection (Infections and infestations) | 2 (2) | 0 (0)
Fungal pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 2 (2)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
H1n1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis b (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis b reactivation (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 5 (5)
Herpes zoster cutaneous disseminated (Infections and infestations) | 1 (1) | 10 (10)
Herpes zoster meningitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster meningoencephalitis (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 11 (11) | 7 (7)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 6 (6) | 2 (2)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 4 (4)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis meningococcal (Infections and infestations) | 1 (1) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (1)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0)
Myelitis (Infections and infestations) | 1 (1) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 3 (3)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 4 (4)
Peritonitis (Infections and infestations) | 0 (0) | 2 (2)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 55 (64) | 41 (46)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 7 (7) | 10 (11)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 15 (15) | 8 (9)
Septic shock (Infections and infestations) | 7 (7) | 5 (5)
Serratia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 2 (2)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Spinal cord abscess (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal scalded skin syndrome (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Immunoglobulins decreased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 8 (8)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angiocentric lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angioimmunoblastic t-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 11 (11)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (14) | 11 (11)
Epstein-barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ewing's sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 3 (3)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 13 (13)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 9 (9)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Peripheral t-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 90 (95) | 70 (71)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Precursor t-lymphoblastic lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 3 (3)
Testicular cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal fistula (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 3 (3) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 3 (3)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vith nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (2)
Drug use disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 12 (12) | 4 (4)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 2 (2)
Renal impairment (Renal and urinary disorders) | 3 (3) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute promyelocytic leukaemia differentiation syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 3 (3)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=922) | Placebo Group (N=924)
Chills (General disorders) | 238 (303) | 117 (134)
Erythema (Skin and subcutaneous tissue disorders) | 304 (422) | 11 (11)
Fatigue (General disorders) | 509 (754) | 341 (496)
Gastrointestinal disorder (Gastrointestinal disorders) | 238 (293) | 185 (235)
Headache (Nervous system disorders) | 304 (391) | 170 (215)
Myalgia (Musculoskeletal and connective tissue disorders) | 485 (718) | 236 (327)
Pain (General disorders) | 757 (1327) | 84 (103)
Pyrexia (General disorders) | 192 (224) | 57 (66)
Swelling (General disorders) | 168 (233) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.